CLINICAL TRIAL: NCT01383629
Title: The Effect of Preoperative Counseling on Patient Fear From Visual Experience During Vitrectomy Surgery Under Regional Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Kenneth Fong, University of Malaya Medical Centre
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UMERC004
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Any Patients Undergoing Vitrectomy Under Local Anaesthesia
Keywords: Vitrectomy; Local anaesthesia; Counselling; Fear; Visual perception
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No counselling (No Intervention): normal preoperative procedures prior to vitrectomy surgery
- Preoperative counselling (Experimental): Counselling to patient about what to expect during vitrectomy surgery under local anaesthesia
  Interventions: Behavioral: Counselling

INTERVENTIONS:
Behavioral: Counselling — Preoperative counselling
  Arms: Preoperative counselling

SUMMARY:
This RCT aims to study the effect of preoperative counselling in reducing patients fear and visual perception during vitrectomy under local anaesthesia.

DETAILED DESCRIPTION:
This was a single-blinded, randomised clinical trial conducted at University of Malaya Medical Centre, Kuala Lumpur, Malaysia, and approved by the Institutional Review Board of the hospital. Patients aged 18-75 years scheduled for vitrectomy under regional anaesthesia were included. Patients who could not understand English, who had psychiatric illness or mental retardation, or who refused to give consent were excluded.

After obtaining informed consent, patients were randomised to two groups: Group A received additional preoperative counseling while Group B did not receive any additional counseling. Both groups received routine preoperative counseling regarding potential risks and benefits of vitrectomy by an ophthalmologist one day prior to the operation.

The information covered during counselling and the method of delivery were standardised for all patients. An ophthalmologist reviewed the patient one day prior to the operation and patients who were randomised to additional counselling were counselled regarding the possible visual perceptions that they might encounter during surgery. These included lights, colours, movements, flashes, instruments and surgeon's hands or face. Twenty four hours after the surgery, another ophthalmologist blinded to the patient randomisation interviewed the patients on their visual perceptions during surgery using a standard questionnaire. Patients were interviewed regarding the types of visual sensations they perceived and if they caused fear to them. Patients were asked to grade their fear based on a visual analogue scale. The fear was graded from 0 to 10, with a score of 0 meaning no fear and a score of 10 being the maximum or extreme fear. At the end of the questionnaire the interviewer was allowed to ask the patient if he or she has received preoperative counselling and if they prefer to be or not to be counselled. Patients were asked to describe in details the images and objects that they saw during the operation. The data were analyzed using SPSS version 17.0.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years scheduled for vitrectomy under regional anaesthesia were included

Exclusion Criteria:

* Patients who could not understand English, who had psychiatric illness or mental retardation, or who refused to give consent were excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Patient fear | 1 week
  Patient fear during surgery is measured on a visual analogue scale

SECONDARY OUTCOMES:
Type of visual perception during vitrectomy surgery under local anaesthesia | 1 week
  Patients visual perception during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Universiy of Malaya Medical Centre, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Tan CS, Mahmood U, O'Brien PD, Beatty S, Kwok AK, Lee VY, Au Eong KG. Visual experiences during vitreous surgery under regional anesthesia: a multicenter study. Am J Ophthalmol. 2005 Dec;140(6):971-975. doi: 10.1016/j.ajo.2005.06.021. PMID 16376638